CLINICAL TRIAL: NCT01683032
Title: A Study on the Effect of Methylphenidate on Creativity of Healthy Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shalvata Mental Health Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: SHA -0011-12
Record Dates: First submitted 2012-08-26; First posted 2012-09-11 (Estimated); Last update posted 2014-11-19 (Estimated); Status verified 2014-11

CONDITIONS: MPH Influence on Creativity
MeSH Terms: interventions — 5,10-dihydro-5-methylphenazine; Methylphenidate

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Experimental: Healthy adults (Experimental): Participants, aged 21-40 years, will be recruited through an advertisement posted at the University of Haifa (including the website of Haifa University).
  Interventions: Drug: MPH

INTERVENTIONS:
Drug: MPH — a capsule containing 20 mg
  Other Names: methylphenidate

SUMMARY:
Creative cognition plays an important role in art, invention and innovation, as well as in everyday life and thus has a significant effect on society as a whole. Research with healthy, normal participants and those with attention deficit hyperactivity disorder indicates a possible inverse relationship between attentional function and creativity. This evidence raises the possibility that Methylphenidate (MPH; Ritalin) could decrease creativity in people using it for cognitive enhancement. However, this question has not been addressed by previous studies. Hence, the present study aims to examine the effect of MPH on creativity in healthy young adults.

DETAILED DESCRIPTION:
Background:

The past decade has seen a rise in the use of prescription stimulants not only by ADHD-diagnosed individual but also by normal healthy individuals for cognitive enhancement. This resulted in a corresponding escalation of illicit use, particularly in college students (confirmed by numerous survey results). In light of this trend, an important issue concerning the effect of cognitive enhancement on the way people think, or what could be called "cognitive style", was raised. Specifically, there has been concern that stimulants might decrease creativity in people using the drugs for cognitive enhancement(.

Creativity has been defined as the ability to produce responses which are both novel (i.e., original, rare and unexpected) and suitable (i.e., adaptive and useful according to the task constrains; ). Many models have been suggested to explain creativity. According to the well established twofold model of creativity, the creative process begins with an associative generation of crudely formed ideas, which is followed by an expansion and exploration of these ideas through a process of evaluation . Since creativity plays an important role in producing novel and useful ideas , it was further speculated that in case of cognitive enhancers continues to be more widely practiced and indeed impair creativity, the effect on society as a whole could be grave The question of whether stimulants might decrease creativity is yet to be elucidated, given that most of previous studies focused on ADHD-diagnosed children, with mixed results; While some of them found that stimulants maintained creativity, others reported it actually worsened the scores on tasks assessing creativity.

Moreover, despite the increase in both illicit and prescribed stimulant use by healthy adults (discussed above) the study by Farah et al.(2009), is so far the only published report investigating stimulant effects on creativity among these individuals. The authors examined the effect of Adderall (a mixture of amphetamine salts) upon creativity, in 16 healthy adults on four tests of creativity, "two tasks requiring divergent thought and two requiring convergent thought (p. 542)." Only performance on the convergent tasks was affected, and the effect depended on baseline performance: in one case enhancing it, particularly for lower-performing individuals, and in the other case enhancing it for the lower-performing and impairing it for higher-performing individuals. This pattern of differential effect of stimulants based on baseline performance, has been noted in other studies of stimulants and cognition and is not unique to creative thought.

Hence, the question of whether stimulants might decrease creativity in healthy adults using the drugs for cognitive enhancement is still open. To best of our knowledge, though MPH is a widely used by healthy normal individuals to enhance cognition, its effect upon creativity of healthy adults has not been studied before. We therefore sought to investigate the effect of MPH upon creativity in healthy adults.

Participants:

The experiment will include a group of 30 healthy adults (male and female). Participants, aged 21-40 years, will be recruited through an advertisement posted at the University of Haifa (including the website of Haifa University).

Screening Phase:

Potential subjects will be required to arrive at the Social and Affective Neuroscience Lab in Haifa University for two visits:

On the first visit, the risks and requirements of this clinical research trial will be explained to each potential subject. Those volunteering to take part will read and sign the Informed Consent Form for participation in the clinical research trial before any trial-related procedures are performed

* Upon obtaining the signed informed consent, inclusion and exclusion criteria will be reviewed to verify the subject's eligibility. Therefore all participants will be interviewed by psychiatrist with the Minimal Structured Clinical Interview for DSM-IV Axis I (SCID-I; First, Gibbons, Spitzer, & Williams, 1995) to exclude those with the presence of lifetime diagnoses of any Axis I disorder.
* In addition, to rule out ADHD, participants will be required to fill in the following questionnaires: conners ADHD Adults Rating-Scale, ASRS v1.1-18 and Wender-Utah self-report rating- scales, Adult ADHD Self-Report Scale (ASRS) Symptom Checklist. Moreover, to rule out any other clinical disorder.
* Each participant will go through a physical examination by a physician and an ECG test to eliminate the risk of previously undiagnosed arrhythmia.

In one of the visits, participants will receive a capsule containing Methylphenidate or placebo (prior to performing the tasks), and in the other visit they will receive a capsule containing placebo. Randomization will be done by the psychiatrist, so that both experimenter and participants are blind to the content of the capsule (The psychiatrist's contact information will be provided in the Informed Consent Form).

MPH dosage will be determined according to participants' body weight: 10 mg in case weight<40 kg; 30 mg in case weight>90 kg; otherwise 20 mg.

ELIGIBILITY:
Inclusion Criteria:

Participants, aged 21-40 years

Exclusion Criteria:

1. People diagnosed with a psychiatric clinical disorder and /or taking psychotropic drugs (whether prescription drugs, herbal extracts or illegal drugs), which may impair their performance in tasks that are used in the study).
2. People for whom there is a contra-indication for consuming Ritalin:

   People who are or were diagnosed with cardiac medical condition, hypertension, liver damage, glaucoma or neurologic disorders (e.g. epilepsy, CVA, parkinson's, Aneurism, brain SOL, MS).
3. Pregnant or nursing women; female participants will be required to report whether they are pregnant, and in case they are, they will not participate.
4. Reported use of drugs at the previous 30 days.

Ages: 21 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2012-10; Primary Completion 2013-05 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
The Alternate Uses Task | 30 min
  This is a standard measure of divergent thinking, whose stimuli and responses are verbal. Subjects will be presented with a list of six common objects (shoe , can, stapler, tire, drinking glass, cardboard box) and will be asked to list as many alternate uses as possible for each object, within a ten minute time limit (the most common everyday use is indicated in parenthesis). Fluency, flexibility and originality will be scored. Original responses will be defined as statistically infrequent responses according to a pretest conducted in our lab

SECONDARY OUTCOMES:
Remote Associates Test (RAT) | 20 min
  The task in a RAT problem is, given three words, to find a fourth word that connects them. (For example, lick, mine, shaker: Answer, salt.) RAT problems require problem solvers to search for distantly related information, and have become a benchmark test of creativity).
The Balloon Analogue Risk Task (BART): | 10 min
  A computerized task of risk-taking behavior in both healthy individuals and in neurological and psychiatric populations. Participants will be able to acquire money by inflating a balloon shown on the computer screen by pressing a key on the keyboard, knowing, however, that the balloon can explode at any time, resulting in the loss of the potential gain. Thus, the participant must balance the potential gain of accruing more money against the potential risk of losing all the money accrued for that balloon.
The Evaluation Task | 10 min
  In the evaluation task participants will be presented with responses of other participants who had performed the AUT previously (with six different items). They will be instructed to rate the general levels of appropriateness of each response and then rate the subcomponents of appropriateness namely, uniqueness, usefulness and deviance by using a 5 points rating scales (ranging from 'not at all' to 'highly' appropriate/unique/useful/deviant).
Torrance Tests for Creative Thinking (TTCT): | 10 min
  the circles subset of the figural part of the TTCT will be used. Participants will be presented with a page of circle. They will be instructed to produce as many different drawings as possible within a time limit of 10 min. Participants will be asked to think of drawings they think no one else could think of. Answers will be scored on fluency, flexibility and originality based on Torrance
Motivation from having an effect | 12 min
  three blocks of trials in which participants respond to colored circles rapidly descanting from the top of the screen. They are then probed from their experience with the task and their motivation to perform it.
visual selection and awareness | 3 min
  a 1-trail task in which participants are oriented to either the inner or outer of two concentric colored circles and then are asked to report the color of both task relevant (oriented) and task irrelevant circles

OTHER OUTCOMES:
Raven Progressive Matrices Test Verbal fluency | 20 min
  1. Verbal fluency: Verbal fluency will be assessed using two items taken from the Controlled Oral Word Association Test (COWAT). In this test the participants are instructed to, during one minute each, generate words beginning with a given letter . All words, except proper nouns and names, are allowed.
  2. Raven Progressive Matrices Test which assesses non-verbal intelligence